CLINICAL TRIAL: NCT03553953
Title: Characterization of Artifacts in the BIS™ EEG Signals in General Anesthesia Patients in Operating Room
Acronym: RAMBAM
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT18003
Record Dates: First submitted 2018-05-31; First posted 2018-06-12 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Anesthesia, General
Keywords: Anesthesia; Bispectral index (BIS™)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients with recording from BIS device: One hundred screened adult patients and no more than 60 valid cases who undergo elective surgery under general anesthesia with recording from the BIS device at the same time and comply with the inclusions criteria
  Interventions: Device: BIS device

INTERVENTIONS:
Device: BIS device — Recording data from BIS device from patients who undergo elective surgery under general anesthesia

SUMMARY:
This is an observational non-invasive study which aims to collect data from patients under general anesthesia in the operating room; this data will then be used for characterization and detection of artifacts that affect the EEG signal.

DETAILED DESCRIPTION:
This observational, non-invasive study will be performed in order to identify the effects of physiological and environmental artifacts on the EEG raw data collected by the BIS™. This study will include 100 screened subjects (not more than 60 valid cases) and will take place in the Department of Anesthesiology at Rambam Health Care Campus. During the study, raw data from the BIS™ will be recorded simultaneously with EMG, EOG and ECG in order to diagnose their effects on the EEG signals as recorded by the BIS™. The raw data will be considered as the main parameters of the study. Additionally, a study coordinator will stay in the operating room during the surgery and will indicate the following parameters -

1. Medical treatment (drug, dosage and time)
2. Changes in hypnotic state (state, time)
3. Any activity that may affect the EEG signals (i.e. electrical and mechanical artifacts from medical devices)
4. Any activity that deviates from the clinical procedure
5. Any adverse events or unusual outcomes From the list above, parameters a, c and d will also be considered as main parameters and parameters and parameters d and e will be considered as safety parameters.

If applicable, BIS™ will be recorded after the surgery, at the PACU, for part of time the subject will be at the PACU or until the subject will be released from the department. The study coordinator/investigator will perform POD assessment at that time. The subject will be considered as valid case even if the data from the recovery room is missing.

Demographic details and medical history will be copied by the study coordinator from the subjects' medical records.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women
* Age >18
* Ability and willingness to participate in the study and sign informed consent form
* Patients that will undergo elective surgery under general anesthesia.

Exclusion Criteria:

* Pregnant women
* Disability or unwillingness to undergo EEG/EMG/ECG measurement
* Subjects with known or suspected sensitivity to adhesive bandage
* Subjects who have sustained CVA or severe head trauma in the last 10 years.
* Subjects with known or suspected electroencephalograph abnormality (e.g. epilepsy or scarring)
* soldiers
* prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include maximum 100 screened adult patients and no more than 60 valid cases who will undergo elective surgery under general anesthesia and who will comply with the inclusions criteria
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2020-08-11 (Actual); Study Completion 2020-08-11 (Actual)

PRIMARY OUTCOMES:
Recording of data that potentially indicates artifacts | 24 hours or less
  The primary objective of the study is to measure and report:
  EMG, EOG and ECG data, each using the respective standard medical device for each parameter; EEG data using the BIS™ device; Environmental events occurring during the same time period (e.g. electrical artifacts)

SECONDARY OUTCOMES:
The effect of demographic and clinical parameters on EEG | week or less
  Generating a database of demographic and clinical data (e.g. level of consciousness, age, gender, BMI, anesthetic agents being used during the study, ASA level, etc.) in order to measure its effect on the EEG data collected with the BIS™.
Immediate post-operative data | week or less
  collect post-operative data in order to assess correlation between EEG data collected with the BIS™ and immediate post-operative delirium (POD)

CONTACTS AND LOCATIONS:
Overall Officials: Aeyal Raz, MD; Ph.D, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No